CLINICAL TRIAL: NCT01700491
Title: Pilot Study: A Non-Inferiority Trial of the Analgesic Effect of Paravertebral Analgesia to Epidural Analgesia for the Management of Post-Operative Pain After Thoracotomy
Brief Title: Pilot Study: Paravertebral Analgesia vs Epidural Analgesia After Thoracotomy
Acronym: ParaEpi
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting and maintenance of blinding necessary for the trial
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Sadeesh Srinathan, MD, Assistant Professor- Department of Thoracic Surgery, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2012:038
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Hypotension
Keywords: Paravertebral Catheter; Epidural Catheter; Analgesia; Hypotension; Analgesia,Epidural; Analgesia,Paravertebral
MeSH Terms: conditions — Hypotension; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Catheter 0.2% ropivacaine (Active Comparator): Patients will receive an infusion of 0.2% ropivacaine at a range of 0-10 mL/hr through an epidural catheter. They will also receive an infusion of saline at a rate of 0-10 mL/hr through a paravertebral catheter.
  Interventions: Drug: Epidural Catheter 0.2% ropivacaine
- Paravertebral Catheter 0.4% ropivacaine (Active Comparator): Patients will receive an infusion of 0.4% ropivacaine at a range of 0-10mL/hr through a paravertebral catheter. They will also receive an infusion of saline at a range of 0-10mL/hr through an epidural catheter.
  Interventions: Drug: Paravertebral Catheter 0.4% ropivacaine

INTERVENTIONS:
Drug: Epidural Catheter 0.2% ropivacaine — 0.2% ropivacaine into epidural space and saline into paravertebral space
  Arms: Epidural Catheter 0.2% ropivacaine
Drug: Paravertebral Catheter 0.4% ropivacaine — 0.4% ropivacaine into paravertebral space and saline into the epidural space
  Arms: Paravertebral Catheter 0.4% ropivacaine

SUMMARY:
Paravertebral analgesia is non-inferior to epidural analgesia for pain control and superior to epidural analgesia in terms of the main complication of hypotension.

DETAILED DESCRIPTION:
There is some evidence that paravertebral analgesia is similar to epidural analgesia in efficacy but superior in maintenance of blood pressure. This is a double blind, randomized control trial comparing paravertebral catheters to epidural catheters for the management of post thoracotomy analgesia. Both groups will undergo placement of a pre-induction epidural catheter as well as a surgically placed paravertebral catheter. Patients will also receive PCA morphine. The primary outcome will be daily morphine use measured in milligrams. The co-primary outcome will be time spent with a systolic blood pressure below 90mmHg. Outcomes will be measured during the first five postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Open thoracotomy
* Age > 18 yo
* Able to use a patient controlled analgesia device

Exclusion Criteria:

* Previous thoracotomy
* Previous spine surgery
* Chronic pain condition
* Ongoing narcotic use
* Prior narcotic abuse
* Active chest infection
* Chest trauma
* Anticoagulation
* Other contraindication to epidural catheter placement
* Allergy to local anesthetic or narcotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Analgesic Effect | At postoperative day 5
  Total cumulative dose of morphine equivalent narcotics.

SECONDARY OUTCOMES:
Hypotension | At postoperative day 5
  Cumulative time in which the systolic blood pressure is below 90mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sadeesh Srinathan, MD, FRCS C-Th, FRCS(C), Principal Investigator — University of Manitoba; Stephen Kowalski, MD, FRCP, Study Chair — University of Manitoba; Rob Brown, MD, FRCP, Study Director — University of Manitoba; Purnima Rao, MD, Study Director — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada